CLINICAL TRIAL: NCT00990548
Title: Family Cardiac Caregiver Investigation to Evaluate Outcomes (FIT-O)
Brief Title: Family Cardiac Caregiver Investigation to Evaluate Outcomes
Acronym: FIT-O
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAE1561; R01HL075101-05A1 (NIH)
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
Keywords: Cardiac Caregivers; Cardiac Patient Clinical Outcomes; Prevention of CVD
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiovascular Service Line patients: Patients admitted to the Cardiovascular Service Line at a major teaching hospital during a consecutive 11-month period.

SUMMARY:
The purpose of the FIT-O study was to estimate the prevalence of having a caregiver (paid and/or informal) among hospitalized cardiac patients by demographic factors such as patient age and race/ethnicity, and to link caregiver status to clinical outcomes following hospitalization. A secondary aim was to collect anonymous family tree data to provide an estimate of the number of first degree family members, their basic demographics, and the distance at which they live from the medical center.

DETAILED DESCRIPTION:
It has been established that cardiac caregivers are a vehicle by which health information can be transmitted, and that caregivers themselves may be at increased CVD risk. Our research evaluated the potential pool and demographic profile of cardiac caregivers as well as the role(s) they play in improving quality of patient care and to enhance adherence to secondary prevention guidelines post discharge. This research also provided important information about targeting educational efforts to specific caregivers to enhance the clinical outcomes of hospitalized coronary patients. The purpose of this study was to estimate the prevalence of caregiving in hospitalized cardiac patients by demographic factors such as patient age and race/ethnicity, and to link caregiving to clinical outcomes in cardiac patients. A secondary aim was to collect family tree data which would allow us to estimate the number of first degree family members, their basic demographics, and the distance at which they live from the medical center in order to determine the feasibility and scope of a targeted preventive intervention. The significance of this research is that it addressed specific challenges outlined in the recent NHLBI strategic plan to develop and evaluate programs to improve patient, provider, and health care system behavior and performance to enhance quality of care and health outcomes, especially in populations that experience a disproportionate disease burden. Unique information was obtained about caregivers as a potential intervention to improve preventive care and health outcomes of patients and families that suffer disproportionate CVD burden. Improved adherence to evidence-based preventive therapies could have a substantial public health benefit.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients admitted to the Cardiovascular Service Line at Columbia University Medical Center/New York-Presbyterian Hospital during a consecutive 11-month period will receive a survey as a routine part of hospital admission.

Exclusion Criteria:

* Inability to read or understand English or Spanish.
* Refusal to complete survey.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiovascular Service Line inpatients at Columbia University Medical Center/New York Presbyterian Hospital during a consecutive 11-month period.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and demographic characteristics of cardiac caregivers among consecutively admitted patients with an acute atherosclerotic coronary event or surgical or catheter-based coronary revascularization procedure. | Upon admission to a major academic teaching hospital
  Cardiac caregivers were classified as either an unpaid family member or friend who assist the patient in complying with medical and lifestyle therapies post-discharge or as a paid professional caregiver. Standardized data were collected on the nature of the tasks the caregiver performs and the caregiver's relationship to the hospitalized patient.

SECONDARY OUTCOMES:
To determine the relation between having or not having a cardiac caregiver and patient clinical outcomes post hospital discharge adjusted for patient demographic characteristics, admitting diagnoses, and co-morbidities. | At admission and 1-year post-hospital discharge

OTHER OUTCOMES:
To collect data regarding the number of family members and their proximity to the hospital to determine the feasibility of an extended family-centered educational and behavioral intervention targeted to family members of patients hospitalized with CVD. | The first 6 months of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lori Mosca, MD, MPH, PhD, Principal Investigator — Columbia University Medical Center/New York-Presbyterian Hosptial
Locations (1):
- Columbia University Medical Center/New York-Presbyterian Hosptial, New York, New York, United States

REFERENCES:
- [Result] Aggarwal B, Liao M, Mosca L. Medication adherence is associated with having a caregiver among cardiac patients. Ann Behav Med. 2013 Oct;46(2):237-42. doi: 10.1007/s12160-013-9492-8. PMID 23536121
- [Result] Mochari-Greenberger H, Mosca M, Aggarwal B, Umann TM, Mosca L. Caregiver status: a simple marker to identify cardiac surgery patients at risk for longer postoperative length of stay, rehospitalization, or death. J Cardiovasc Nurs. 2014 Jan-Feb;29(1):12-9. doi: 10.1097/JCN.0b013e318274d19b. PMID 23321779
- [Result] Hammond G, Mochari-Greenberger H, Liao M, Mosca L. Effect of gender, caregiver, on cholesterol control and statin use for secondary prevention among hospitalized patients with coronary heart disease. Am J Cardiol. 2012 Dec 1;110(11):1613-8. doi: 10.1016/j.amjcard.2012.07.028. Epub 2012 Aug 15. PMID 22901971
- [Result] Mosca L, Aggarwal B, Mochari-Greenberger H, Liao M, Blair J, Cheng B, Comellas M, Rehm L, Suero-Tejeda N, Umann T. Association between having a caregiver and clinical outcomes 1 year after hospitalization for cardiovascular disease. Am J Cardiol. 2012 Jan 1;109(1):135-9. doi: 10.1016/j.amjcard.2011.07.072. Epub 2011 Sep 29. PMID 21962999
- [Result] Mosca L, Mochari-Greenberger H, Aggarwal B, Liao M, Suero-Tejeda N, Comellas M, Rehm L, Umann TM, Mehran R. Patterns of caregiving among patients hospitalized with cardiovascular disease. J Cardiovasc Nurs. 2011 Jul-Aug;26(4):305-11. doi: 10.1097/JCN.0b013e3181f34bb3. PMID 21330929
- [Result] Villanueva C, Aggarwal B. The association between neighborhood socioeconomic status and clinical outcomes among patients 1 year after hospitalization for cardiovascular disease. J Community Health. 2013 Aug;38(4):690-7. doi: 10.1007/s10900-013-9666-0. PMID 23468321
- [Result] Blair J, Volpe M, Aggarwal B. Challenges, needs, and experiences of recently hospitalized cardiac patients and their informal caregivers. J Cardiovasc Nurs. 2014 Jan-Feb;29(1):29-37. doi: 10.1097/JCN.0b013e3182784123. PMID 23416934